CLINICAL TRIAL: NCT06096766
Title: Study on the Correlation Between Ovarian Function and Serum Biomarkers
Brief Title: The Correlation Between Ovarian Function and Serum Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Shi Yun (Other)
Responsible Party: Sponsor-Investigator, Shi Yun, Sponsor-Investigator, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Other Study IDs: 2023DZMEC-489
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Premature Ovarian Insufficiency; Diminished Ovarian Reserve; Biomarker; Copper; Ceruloplasmin; Aging
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diminished Ovarian Reserve Group: women with DOR
  Interventions: Diagnostic Test: blood test
- Premature Ovarian Insufficiency Group (POI): women with premature ovarian insufficiency
  Interventions: Diagnostic Test: blood test
- Control Group: women with normal menstruation and levels of sex hormones
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — Detection of serum levels of copper ions, iron ions, ceruloplasmin (CP), CuZn SOD, malondialdehyde (MDA), etc. Blood samples will be retained from the rest samples for sex hormones samples for testing sex hormones, which don't increase times of blood collection.

SUMMARY:
The goal of this observational study is to find differences in serum biomarkers between ovarian function and normal individuals.

DETAILED DESCRIPTION:
Collect the serum of the observation group and control group volunteers, and measure the levels of copper ions, iron ions, ceruloplasmin (CP), CuZn SOD, malondialdehyde (MDA), etc. in the serum.

ELIGIBILITY:
Inclusion Criteria:

1. The selection criteria for healthy individuals are follows.

   * women aged 18-45.

     * Basic FSH<10IU/L, and AMH is within the normal range.

       * Regular menstruation.

         * Agree and sign an informed consent form.
2. The selection criteria for DOR patients are follows.

   * women aged 18-45.

     * For two consecutive menstrual cycles, 25 ≥ basal FSH ≥ 10IU/L or AMH<1.1ng/ml.

       * Agree and sign an informed consent form.
3. Selection criteria for POI patients are follows.

   * 18 ≤ females aged <40 years old.

     * Two consecutive menstrual cycles with basal FSH>25IU/L or AMH<1.1ng/ml.

       * Agree and sign an informed consent form.

Exclusion Criteria:

1. Patients with congenital gonadal developmental abnormalities or a family history similar to "early menopause".
2. Patients with acquired organic lesions or decreased ovarian function caused by ovarian surgery.
3. Patients who have undergone artificial cycle therapy with Western medicine or other endocrine treatments within the past three months.
4. Patients with severe primary diseases and mental disorders such as crdiovascular, cerebrovascular, liver, kidney, and hematopoietic system.
5. Patients during lactation or pregnancy.
6. Patients who are allergic to the drugs used in this study or have a history of allergic reactions to traditional Chinese medicine.

Those who meet any of the above 5 criteria for DOR and POI will be excluded and not included in this study. The exclusion criteria for healthy subjects are as (1), (3), (4), and (5).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological sex
Study Population: Visited the gynecology clinic of Dongzhimen Hospital from November 2023 to October 2024. Upon examination of sexual hormones or AMH, it was considered that patients with Diminished Ovarian Reserve (DOR), premature ovarian insufficiency (POI), and healthy individuals had decreased ovarian reserve function.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-11-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
copper | On the 2~4th day of menstruation (amenorrhea patients on the enrolled week)
  the level of copper in blood sample
Iron ion | On the 2~4th day of menstruation (amenorrhea patients on the enrolled week)
  the level of Iron ion in blood sample
ceruloplasmin, CP | On the 2~4th day of menstruation (amenorrhea patientson the enrolled week)
  the level of ceruloplasmin in blood sample
CuZn-Superoxide Dismutase, CuZn-SOD/SOD1 | On the 2~4th day of menstruation (amenorrhea patients on the enrolled week)
  the level of CuZn-SOD/SOD1 in blood sample
Malondialdehyde，MDA | On the 2~4th day of menstruation (amenorrhea patients on the enrolled week)
  the level of MDA in blood sample

SECONDARY OUTCOMES:
other relative biomarkers about copper/iron metabolism and oxidative stress | On the 2~4th day of menstruation (amenorrhea patients on the enrolled week)
  depending on the results of the five biomarkers above

CONTACTS AND LOCATIONS:
Overall Officials: Yun Shi, PhD, Study Director — Dongzhimen Hospital of Beijing University of Chinese Medicine; Ke Xu, Master, Principal Investigator — Dongzhimen Hospital of Beijing University of Chinese Medicine; Jing Y Shao, Master, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Xuan kai Cai, Master, Study Chair — Shenzhen Bao'an Authentic TCM Therapy Hospital; Qin Y Liu, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Xi Y Li, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Fei Yan, Master, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China

IPD SHARING:
Plan to Share IPD: No